CLINICAL TRIAL: NCT03562481
Title: Pilot Study: Comparison of Buffered 1% vs. Unbuffered 2% Lidocaine in Pediatric Subjects; Clinical Outcomes
Brief Title: Clinical Trial Comparing Effectiveness of Buffered Versus Unbuffered Local Anesthetic in Children Ages 10-12 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 16-3106
Record Dates: First submitted 2018-06-05; First posted 2018-06-19 (Actual); Results first posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-02

CONDITIONS: Anesthesia, Local; Pain
Keywords: Healthy pediatric volunteers
MeSH Terms: conditions — Pain | interventions — Epinephrine; Lidocaine

STUDY DESIGN:
Intervention Model Description: Study subjects will serve as their own controls in this crossover AB/BA study design which is uniform within sequences (groups, i.e. AB/BA, of order of drug formulation administration), uniform within periods (equal time between administration of alternating drug formulations), and balanced (equal number of subjects within each study arm).
  The randomization will be performed to the type of drug given first, using a balanced randomization (half subjects buffered, half unbuffered) implemented with SAS software routines. During the first session, each subject will receive an IAN block with the first randomly assigned anesthetic formulation using the Halstead technique. At least a week later, substantially longer than the elimination half-life of the drug lidocaine (1.5-2hr), local anesthetic injections will be done using the alternate local anesthetic formulation.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Buffered Anesthetic, then Unbuffered Anesthetic (Experimental): Subjects randomized to Buffered Anesthetic, then Unbuffered Anesthetic will first receive an injection with 1% Buffered Lidocaine 1:100,000 Epinephrine. After one week minimum washout period, subjects will then receive an injection with 2% Unbuffered Lidocaine 1:100,000 Epinephrine.
  Interventions: Drug: 1% Buffered Lidocaine 1:100,000 Epinephrine; Drug: 2% Unbuffered Lidocaine 1:100,000 Epinephrine
- Unbuffered Anesthetic, then Buffered Anesthetic (Experimental): Subjects randomized to Unbuffered Anesthetic, then Buffered Anesthetic will first receive an injection with 2% Unbuffered Lidocaine 1:100,000 Epinephrine. After one week minimum washout period, subjects will then receive an injection with 1% Buffered Lidocaine 1:100,000 Epinephrine.
  Interventions: Drug: 1% Buffered Lidocaine 1:100,000 Epinephrine; Drug: 2% Unbuffered Lidocaine 1:100,000 Epinephrine

INTERVENTIONS:
Drug: 1% Buffered Lidocaine 1:100,000 Epinephrine — A single IAN block with 3cc 1% Buffered Lidocaine (30mg) 1:100,000 Epinephrine using the Halstead technique.
  Other Names: Xylocaine
Drug: 2% Unbuffered Lidocaine 1:100,000 Epinephrine — A single IAN block with 3cc 2% Unbuffered Lidocaine (60mg) 1:100,000 Epinephrine using the Halstead technique.
  Other Names: Xylocaine

SUMMARY:
Local anesthesia is an integral part of clinical pediatric dental practice, but it has challenges. It can be uncomfortable for children, and the risk of adverse events limits how much is used. Some evidence suggests benefits of buffering local anesthetics including equal effect with less pain on injection. These findings have not been replicated and validated among pediatric populations, creating a gap in the knowledge base. To address this knowledge gap and contribute to the evidence base on safety and efficacy of local anesthesia in pediatric dentistry, this investigation proposes to compare the anesthetic effects of buffered 1% lidocaine with those of unbuffered 2%, among children.

The specific aims of this investigation are to determine differences between buffered 1% and unbuffered 2% lidocaine (both with 1:100,000 epinephrine) used for inferior alveolar nerve block (IAN) anesthesia, in the following domains:

1. Pain experience on injection, time to onset following the administration, and time to recovery [subjective]
2. Blood lidocaine levels 15 minutes following the administration and duration of pulpal anesthesia [objective]

Null Hypotheses:

1. No difference exists in anesthetic effectiveness for pulpal anesthesia after intraoral IAN block between buffered 1% Lidocaine with 1:100,000 epinephrine as compared to unbuffered 2% Lidocaine with 1:100,000 epinephrine.
2. No differences exist in peak blood lidocaine levels, pain on injection, time to lip numbness, and duration of anesthesia between the two drug formulations.

Randomized subjects will be injected orally for bottom jaw anesthesia, with 3cc of buffered 1% lidocaine (30mg) 1:100,000 epinephrine or 3cc unbuffered of 2% lidocaine (60mg) 1:100,000 epinephrine. The injectable volume of the buffered formulation will include 0.3cc of 8.4% sodium bicarbonate.

One faculty member in the Department of Pediatric Dentistry at the University of North Carolina (UNC) School of Dentistry will administer the drugs in the Pediatric Dentistry clinic. The same clinician will administer injection to the same subjects at both visits. Clinicians and subjects will not know which drug formulation is given at which appointment.

A clinician will measure the level of discomfort on injection, how long it takes for the lip to be numb, how long it takes for the first molar tooth in that area to be numb, how long it takes the local anesthetic to wear off, and how much of the anesthetic is in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-12 years
* American Society of Anesthesiologists (ASA) Class I (Healthy)
* Body Weight: the Interquartile Range (IQR) 33-60Kg for subject ages
* Have ability to speak and read English
* Willingness to participate in two sessions
* No history of adverse reaction to dental anesthetic
* Have bilateral, disease/symptom-free mandibular first molars present

Exclusion Criteria:

* Allergy to lidocaine class of anesthetic drugs
* Local anesthetic drug use in past week
* Current symptomatic teeth or oral mucosa
* ASA II or above (including asthma)

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Y Lee, DDS,MPH,PhD, Principal Investigator — UNC-Chapel Hill School of Dentistry, Pediatric Dentistry
Locations (1):
- UNC School of Dentistry, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB) and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: 9 to 36 months following publication
Access Criteria: Investigators who propose to use the data must have approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB) and must execute a data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Unbuffered Anesthetic, Then Buffered Anesthetic: Subjects randomized to Unbuffered Anesthetic, then Buffered Anesthetic will first receive an injection with 2% Unbuffered Lidocaine 1:100,000 Epinephrine. 1% After one week minimum washout period, subjects will then receive an injection with Buffered Lidocaine 1:100,000 Epinephrine.
- Sequence 2: Buffered Anesthetic, Then Unbuffered Anesthetic: Subjects randomized to Buffered Anesthetic, then Unbuffered Anesthetic will first receive an injection with 1% Buffered Lidocaine 1:100,000 Epinephrine. After one week minimum washout period, subjects will then receive an injection with 2% Unbuffered Lidocaine 1:100,000 Epinephrine.
Period: First Intervention
Arm/Group | Sequence 1: Unbuffered Anesthetic, Then Buffered Anesthetic | Sequence 2: Buffered Anesthetic, Then Unbuffered Anesthetic
Started | 12 | 14
Completed | 11 | 14
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Washout
Arm/Group | Sequence 1: Unbuffered Anesthetic, Then Buffered Anesthetic | Sequence 2: Buffered Anesthetic, Then Unbuffered Anesthetic
Started | 11 | 14
Completed | 11 | 14
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Sequence 1: Unbuffered Anesthetic, Then Buffered Anesthetic | Sequence 2: Buffered Anesthetic, Then Unbuffered Anesthetic
Started | 11 | 14
Completed | 11 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence 1: Unbuffered Anesthetic, Then Buffered Anesthetic: Subjects randomized to Unbuffered Anesthetic, then Buffered Anesthetic will first receive an injection with 2% Unbuffered Lidocaine 1:100,000 Epinephrine. After one week minimum washout period, subjects will then receive an injection with 1% Buffered Lidocaine 1:100,000 Epinephrine.
- Total: Total of all reporting groups
Arm/Group | Sequence 1: Unbuffered Anesthetic, Then Buffered Anesthetic | Sequence 2: Buffered Anesthetic, Then Unbuffered Anesthetic | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.5 (0.5) | 10.9 (0.9) | 11.2 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 8 | 5 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Black | 4 | 1 | 5
  White | 7 | 12 | 19
  Other | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 14 | 26
Response to Cold Testing [Count of Participants; unit: Participants]
  Negative Response to Cold Testing at Baseline | 2 | 4 | 6
  Positive Response to Cold Testing at Baseline | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean Pain Scores Following Injection
Description: Perceived pain on injection, self-reported verbally using a Likert scale from 1-10, with lower numbers corresponding to less pain (1 = "no pain," 10 = "worst pain imaginable"). Lower scores reflect a lesser degree of pain.
Time Frame: Within 10 minutes of injection
Population: One participant did not complete the second intervention and was excluded from the data analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Buffered Anesthetic: Subjects being administered the Buffered Anesthetic received an injection with 3cc 1% Buffered Lidocaine 1:100,000 Epinephrine. for a single IAN block using the Halstead technique.
  1% Buffered Lidocaine 1:100,000 Epinephrine: A single IAN block with 3cc 1% Buffered Lidocaine (30mg) 1:100,000 Epinephrine using the Halstead technique.
- Unbuffered Anesthetic: Subjects being administered the Unbuffered Anesthetic received an injection with 3cc of 2% Unbuffered Lidocaine with 1:100,000 Epinephrine for a single IAN block using the Halstead technique.
  2% Unbuffered Lidocaine 1:100,000 Epinephrine: A single IAN block with 3cc 2% Unbuffered Lidocaine (60mg) 1:100,000 Epinephrine using the Halstead technique.
Arm/Group | Buffered Anesthetic | Unbuffered Anesthetic
Number analyzed (Participants) | 25 | 25
score on a scale | 3.0 (1.9) | 3.3 (1.5)
Statistical Analysis 1: Comparison: Buffered Anesthetic vs Unbuffered Anesthetic; Test type: Equivalence — Analysis of variance for a 2x2 crossover study implemented using the pkcross routine of Stata 16.1, accounting of sequence and period effects; p = 0.38, ANOVA — The threshold for statistical significance p<0.05; Analysis of variance for a 2x2 crossover study implemented using the pkcross routine of Stata 16.1, accounting of sequence and period effects; F statistic = 0.80

2. Primary Outcome: Mean Time to Lower Lip Numbness Following Injection
Description: Time in minutes beginning immediately following injection to patient-reported lip numbness
Time Frame: Up to 30 minutes following injection
Population: One participant did not complete the second intervention and was excluded from the data analysis.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Buffered Anesthetic: Subjects randomized to Buffered Anesthetic, then Unbuffered Anesthetic will first receive an injection with 1% Buffered Lidocaine 1:100,000 Epinephrine. After one week minimum washout period, subjects will then receive an injection with 2% Unbuffered Lidocaine 1:100,000 Epinephrine.
  1% Buffered Lidocaine 1:100,000 Epinephrine: A single IAN block with 3cc 1% Buffered Lidocaine (30mg) 1:100,000 Epinephrine using the Halstead technique.
- Unbuffered Anesthetic: Subjects randomized to Unbuffered Anesthetic, then Buffered Anesthetic will first receive an injection with 2% Unbuffered Lidocaine 1:100,000 Epinephrine. After one week minimum washout period, subjects will then receive an injection with 1% Buffered Lidocaine 1:100,000 Epinephrine.
  2% Unbuffered Lidocaine 1:100,000 Epinephrine: A single IAN block with 3cc 2% Unbuffered Lidocaine (60mg) 1:100,000 Epinephrine using the Halstead technique.
Arm/Group | Buffered Anesthetic | Unbuffered Anesthetic
Number analyzed (Participants) | 25 | 25
minutes | 3.4 (1.3) | 4.4 (3.7)
Statistical Analysis 1: Comparison: Buffered Anesthetic vs Unbuffered Anesthetic; Analysis of variance for 2x2 crossover study using the pkcross routine of Stata 16.1 and accounting for sequence and period effects; Test type: Equivalence — Equivalence was defined as a non-statistically significant difference; p = 0.28, ANOVA — The threshold for statistical significance p<0.05; F statistic = 1.21

3. Primary Outcome: Average Serum Lidocaine Concentration at 15 Minutes Post Injection
Description: Blood Lidocaine Level (mcg/mL) as measured in 10cc venous blood, taken 15 minutes following injection. Blood assayed for serum lidocaine levels with a Sciex TripleTOF liquid chromatography- mass spectrometry (LC-MS) equipped with a C18 Hypersil (10mm x 2.1mm, 3.0μm).
Time Frame: One blood draw taken 15 minutes following injection
Population: One participant did not complete the second intervention and was excluded from the data analysis.
Measure: Mean (Standard Deviation); unit: mcg/ml
Arm/Group | Buffered Anesthetic | Unbuffered Anesthetic
Number analyzed (Participants) | 25 | 25
mcg/ml | 243.5 (127.9) | 600.2 (497.0)
Statistical Analysis 1: Comparison: Buffered Anesthetic vs Unbuffered Anesthetic; Analysis of variance for 2x2 crossover study using the pkcross routine of Stata 16.1 adjusting for perio and sequence effects; Test type: Equivalence — Equivalence was defined based on statistical significance in the cross-over ANOVA; p = 0.003, ANOVA — This is adjusted for period and sequence effects and is statistically significant at the p<0.05 level; F statistic = 11.1

4. Primary Outcome: Mean Time to Baseline Lip Sensation
Description: Response in minutes from injection to when lip is no longer numb, as self reported by patient.
Time Frame: Within 24 hours following injection
Population: One participant did not complete the second intervention and was excluded from the data analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Buffered Anesthetic | Unbuffered Anesthetic
Number analyzed (Participants) | 25 | 25
minutes | 218 (59.6) | 241 (91.4)
Statistical Analysis 1: Comparison: Buffered Anesthetic vs Unbuffered Anesthetic; Test type: Equivalence — Equivalence was determined based on the statistical significance of the Wilcoxon signed-rank test; p = 0.33, Sign test — The threshold for statistical significance p<0.05; Wilcoxon signed-rank test; Z score = -0.996

5. Primary Outcome: Number of Participants Who Respond to Cold Stimulus (Positive/Negative) Prior to Injection
Description: Response to experiencing sensation to cold stimulus on permanent molar tooth prior to injection
Time Frame: 5 minutes prior to injection
Population: One participant did not complete the second intervention and was excluded from the data analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Buffered Anesthetic: 1% Buffered Lidocaine 1:100,000 Epinephrine: A single IAN block with 3cc 1% Buffered Lidocaine (30mg) 1:100,000 Epinephrine using the Halstead technique.
- Unbuffered Anesthetic: 2% Unbuffered Lidocaine 1:100,000 Epinephrine: A single IAN block with 3cc 2% Unbuffered Lidocaine (60mg) 1:100,000 Epinephrine using the Halstead technique.
Arm/Group | Buffered Anesthetic | Unbuffered Anesthetic
Number analyzed (Participants) | 25 | 25
Participants
  Negative Response to Cold Testing at Baseline | 6 | 2
  Positive Response to Cold Testing at Baseline | 19 | 23
Statistical Analysis 1: Comparison: Buffered Anesthetic; Test type: Equivalence — Equivalence was determined based on the statistical significance of the chi square test; p = 0.37, Chi-squared — The threshold for statistical significance p<0.05; Chi-square test = 0.81

6. Primary Outcome: Number of Participants Who Respond to Cold Stimulus (Positive/Negative) 30 Minutes Following Injection
Description: Response to experiencing sensation to cold stimulus on permanent molar tooth 30 minutes following injection
Time Frame: 30 minutes following injection
Population: One participant did not complete the second intervention and was excluded from the data analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Buffered Anesthetic | Unbuffered Anesthetic
Number analyzed (Participants) | 25 | 25
Participants
  Negative Response to Cold Testing | 17 | 18
  Positive Response to Cold Testing | 8 | 7
Statistical Analysis 1: Comparison: Buffered Anesthetic vs Unbuffered Anesthetic; Stuart-Maxwell test of marginal homogeneity implemented with the symmetry routine in Stata 16.1; Test type: Equivalence — Equivalence was defined based on statistical significance in the symmetry test; p = 0.65, Sruart-Maxwell symmetry test — The threshold for statistical significance p<0.05; Chi-square test = 0.20

7. Primary Outcome: Number of Participants Who Respond to Cold Stimulus (Positive/Negative) 60 Minutes Following Injection
Description: Response to experiencing sensation to cold stimulus on permanent molar tooth 60 minutes following injection
Time Frame: 60 minutes following injection
Population: One participant did not complete the second intervention and was excluded from the data analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Buffered Anesthetic | Unbuffered Anesthetic
Number analyzed (Participants) | 25 | 25
Participants
  Negative Response to Cold Testing | 17 | 18
  Positive Response to Cold Testing | 8 | 7
Statistical Analysis 1: Comparison: Buffered Anesthetic vs Unbuffered Anesthetic; Test of symmetry or marginal homogeneity (Stuart-Maxwell) implemented with the symmetry routine in Stata 16.1; Test type: Equivalence — Equivalence was defined based on significance in the symmetry test; p = 0.71, Sruart-Maxwell symmetry test — The threshold for statistical significance p<0.05; Chi-square test = 0.14

8. Primary Outcome: Number of Participants Who Respond to Cold Stimulus (Positive/Negative) 90 Minutes Following Injection
Description: Response to experiencing sensation to cold stimulus on permanent molar tooth 90 minutes following injection
Time Frame: 90 minutes following injection
Population: One participant did not complete the second intervention and was excluded from the data analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Buffered Anesthetic | Unbuffered Anesthetic
Number analyzed (Participants) | 25 | 25
Participants
  Negative Response to Cold Testing | 15 | 18
  Positive Response to Cold Testing | 10 | 7
Statistical Analysis 1: Comparison: Buffered Anesthetic vs Unbuffered Anesthetic; Test of symmetry (marginal homogeneity, Stuart-Maxwell) implemented using the symmetry routine in Stata 16.1; Test type: Equivalence — Equivalence was defined based on statistical significance in the symmetry test; p = 0.32, Sruart-Maxwell symmetry test — The threshold for statistical significance p<0.05; Chi-square test = 1.00

9. Primary Outcome: Number of Participants Who Respond to Cold Stimulus (Positive/Negative) 120 Minutes Following Injection
Description: Response to experiencing sensation to cold stimulus on permanent molar tooth 120 minutes following injection
Time Frame: 120 minutes following injection
Population: One participant did not complete the second intervention and was excluded from the data analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Buffered Anesthetic | Unbuffered Anesthetic
Number analyzed (Participants) | 25 | 25
Participants
  Negative Response to Cold Testing | 13 | 19
  Positive Response to Cold Testing | 12 | 6
Statistical Analysis 1: Comparison: Buffered Anesthetic vs Unbuffered Anesthetic; Test of symmetry (marginal homogeneity, Stuart-Maxwell) implemented using the symmetry routine in Stata 16.1; Test type: Equivalence — Equivalence was defined based on the statistical significance of the symmetry test; p = 0.26, Sruart-Maxwell symmetry test; Chi-square test = 1.29

ADVERSE EVENTS:
Time Frame: Following randomization through the end of Intervention 2, up to approximately 8 weeks.
Arm/Group | Buffered Anesthetic | Unbuffered Anesthetic
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 0/25 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT03562481/Prot_SAP_000.pdf